CLINICAL TRIAL: NCT00727701
Title: Does Use of a Wound After-care Summary for Patients With a History of Venous Ulcers Lower Recurrence Rate?
Brief Title: Study of Individualized Wound Prevention Instruction to Prevent Venous Ulcer Development
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study delayed for over a year by research shutdown at Seattle VA and other issues. Study designer moved to Ann Arbor in the interim, so the study was closed.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Reiber, Gayle - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-246
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Varicose Ulcer
Keywords: varicose ulcer; veteran; recurrence; aftercare
MeSH Terms: conditions — Varicose Ulcer; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Will receive usual wound prevention care, aftercare summaries, and regular surveillance.
  Interventions: Behavioral: Aftercare summary
- 2 (No Intervention): Will receive usual wound prevention and surveillance only.
- 3 (No Intervention): Will receive usual wound prevention only.

INTERVENTIONS:
Behavioral: Aftercare summary — A personalized, targeted set of self-care instructions for venous ulcer prevention, including a graphical depiction of patient adherence to self-care goals.
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether individualized wound prevention instructions will lengthen the ulcer-free period in veterans with recently healed venous ulcers.

DETAILED DESCRIPTION:
Venous ulcer disease is the most common form of lower extremity ulcer, and treatment requires months to years of costly intervention. Preventing venous ulcers from recurring is ideal, however, healing time is variable, possibly due to inadequate patient/clinician communication and surveillance. An aftercare summary is a detailed set of self-care instructions designed to help patients understand and influence preventative factors under their control. They have successfully been used in patients with cardiac disease and are currently being tested to help prevent diabetic foot ulcers. We propose the use of an aftercare summary to help prevent ulcer recurrence in veterans with recently healed venous ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed venous ulcer (ICD-9: 454.0, 454.2, 459.11, 459.13, 459.31, 459.33);
* Documented healing of all lower extremity ulcers;
* Ankle-brachial index (ABI) > 0.8 to rule out arterial insufficiency

Exclusion Criteria:

* Unwilling or unable to sign informed consent;
* No plans to seek care at VA Puget Sound within 6 months;
* Limbs with ulcers or threatened viability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Ulcer-free survival period | Telephone call every 2 weeks, on-site visit quarterly (depends on study arm)

SECONDARY OUTCOMES:
Change in quality of life | Telephone call every 2 weeks, on-site visit at 2.5 and 5 months.
Change in satisfaction with care | Telephone call every 2 weeks, on-site visit at 2.5 and 5 months.
Adherence with self-management goals | Telephone call every 2 weeks, on-site visit at 2.5 and 5 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gayle E. Reiber, MPH PhD, Principal Investigator — VA Puget Sound Health Care System, Seattle
Locations (1):
- VA Puget Sound Health Care System, Seattle, Seattle, Washington, United States